CLINICAL TRIAL: NCT04153266
Title: Development of an Oral Epithelial Dysplasia Informational Needs Questionnaire
Brief Title: Oral Epithelial Dysplasia Informational Needs Questionnaire
Acronym: ODIN-Q
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0203
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Oral Epithelial Dysplasia; Precancerous Conditions; Precancerous Lesions; Oral Lichen Planus; Oral Leukoplakia; Oral Leukoplakia of Tongue; Oral Leukoplakia of Lips; Oral Leukoplakia of Gingiva; Oral Erythroplakia; Chronic Hyperplastic Candidosis; Oral Submucous Fibrosis; Oral Submucosal Fibrosis, Including of Tongue; Oral Disease; Dental Diseases; Dysplasia; Information Seeking Behavior; Patient Preference; Information Needs; Health Behavior; Quality of Life; Preference, Patient; Patient Satisfaction; Patient Engagement; Patient Participation
Keywords: oral epithelial dysplasia; Precancerous Conditions; Precancerous Lesions; Information Seeking Behavior; Patient Preference; Oral Disease; Dental Diseases; Dysplasia; Quality of Life; Patient Satisfaction; Patient Participation; information needs; patient education; patient information leaflet
MeSH Terms: conditions — Precancerous Conditions; Lichen Planus, Oral; Leukoplakia, Oral; Oral Submucous Fibrosis; Mouth Diseases; Stomatognathic Diseases; Information Seeking Behavior; Patient Preference; Health Behavior; Patient Satisfaction; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with oral epithelial dysplasia: INCLUSION CRITERIA
  These include:
  * Adults aged 18 or above at the time of the screening visit.
  * Good command of English language both written and spoken [this is necessary as questionnaires are in English and cannot be translated unless through a cross-cultural validation study].
  * Being able to consent.
  * Diagnosed with OED as per current standard diagnostic criteria.
  * No concurrent malignancy in the head and neck or elsewhere.
  Interventions: Other: No intervention is planned for this study

INTERVENTIONS:
Other: No intervention is planned for this study — No intervention was/is planned for this study. The study is questionnaire-based (observational).

SUMMARY:
Background: Oral epithelial dysplasia (OED) is a condition with an increased risk of oral cancer. Due to the current changes in the factors associated with these diseases (because of human papillomavirus), it is expected that those who have no history of smoking or alcohol, young (<50 years old), and white male would be commonly affected. Those individuals require a higher need for information, preferred a more active role in decision-making, and have a longer lifespan than older individuals. There remain no detailed studies of whether the informational needs delivered to patients with OED met their needs or indeed what information such patient may wish. A few tools are available to evaluate the IN of patients with head and neck disorders. However, the items of these instruments were dedicated to a particular disease (e.g. cancer) and hence are not applicable to be used for OED.

Project aims: To evaluate the psychometric properties of the Oral Epithelial Dysplasia Informational Needs Questionnaire (ODIN-Q), developed and revised in the preliminary work for the proposed study, in a cohort of patients with OED.

Timescale: 19 months.

Clinical significance: This questionnaire can be useful in clinical practice. It could help to meet the patient's information needs and plan educational interventions for those showing unmet needs.

DETAILED DESCRIPTION:
Oral epithelial dysplasia (OED) is a disease associated with an increased risk of oral cancer between 6% and 36% compared to disease-free individuals. In the United Kingdom, oral cancer is among the 15 most common cancers, with approximately 6,000 new cases per year and these numbers are expected to rise in the few coming years.

Research showed the importance of patient education and the provision of information in shared-decision making and management of chronic and cancer-linked disease such as perhaps OED. However, patients may not be satisfied with the information provided by healthcare professionals, despite the extensive nature of the information provided. Having unmet informational needs may associate with higher anxiety levels which in turn could affect the patient's well-being and cooperation with the treatment provided.

Avoiding these undesirable health outcomes requires the delivery of tailored and patient-centred care that provides information based on what patients truly need and prefer. One increasingly common method to do so is to obtain this information by informational needs questionnaires. These questionnaires have been developed for other medical conditions including chronic diseases and some cancers, but none of these is known to be appropriate to use for OED specifically. Hence, a specific tool to determine the informational needs and preferences of patients with OED may help to achieve these objectives effectively. The data collected by this tool may help to acknowledge the impact of the illness on physical and psychological well-being. Furthermore, this data could be used to produce a source of OED information (such as a patient information leaflet) that reflects the IN of this patient population.

In the preliminary work for this study, the Oral Epithelial Dysplasia Informational Needs Questionnaire (ODIN-Q) was developed by adopting existing valid and reliable instruments that explore the information need of patients with potentially malignant disease elsewhere in the body, using experts input. The questions were then formulated and tested for content validity by clinicians (n=12) and patients (n=5), with unclear, irrelevant, redundant, and unacceptable items omitted. The final 35-item ODIN-Q includes two scales: (1) amount of information already received (too much, enough, not enough and none) and (2) degree of importance of the information (very, yes, not very, not at all).

Thus, the objectives of this study are to (1) test the newly developed ODIN-Q in a cohort of patients with OED; (2) to investigate the correlations between patients' informational needs and both of psychological variables (e.g. anxiety and depression) and quality of life; and (3) to develop and a Patient Information Leaflet (PIL) for OED based on patients' needs and preferences.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or above at the time of the screening visit.
* Good command of English language both written and spoken.
* Being able to consent.
* Diagnosed with OED by histopathological examination as per the 2017 classification of head and neck tumours by the World Health Organization.
* No concurrent malignancy in the head and neck or elsewhere.

Exclusion Criteria:

* Individuals under 18 years old.
* Unable to speak and read English.
* Concurrent malignancy in the head and neck or elsewhere.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients diagnosed with OED as per current standard diagnostic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
ODIN-Q validation | 14 months
  To evaluate the psychometric properties of the Oral Epithelial Dysplasia Informational Needs Questionnaire (ODIN-Q), developed and revised in the preliminary work for the proposed study, in a cohort of patients with OED (Phase 1).

SECONDARY OUTCOMES:
Correlations between information needs and other variables measured in the study | 14 months
  To investigate the correlation between psychological variables (e.g. anxiety and depression), quality of life (QoL) and information needs by analysis of the data collected by ODIN-Q, Krantz Health Opinion Survey, Hospital Anxiety and Depression Scale, Modified Dental Anxiety Scale and the Oral Health Impact Profile-14 (phase 1).
Develop a patient information leaflet about oral epithelial dysplasia | 14 months
  To develop and assess the satisfaction with a patient information leaflet [PIL] about OED (phase 2).

CONTACTS AND LOCATIONS:
Locations (1):
- University college london hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alsoghier A, Ni Riordain R, Fedele S, Porter S. Web-based information on oral dysplasia and precancer of the mouth - Quality and readability. Oral Oncol. 2018 Jul;82:69-74. doi: 10.1016/j.oraloncology.2018.05.003. Epub 2018 May 17. PMID 29909904
- See also: Preparatory work to inform the current study — https://www.ncbi.nlm.nih.gov/pubmed/?term=Web-based+information+on+oral+dysplasia+and+precancer+of+the+mouth+-+Quality+and+readability